CLINICAL TRIAL: NCT00413127
Title: Perioperative Protective Effects of Lidocaine - Clinical Study on the Route and Timing of Administration
Brief Title: Perioperative Protective Effects of Lidocaine
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Less patients than expected for inclusion, therefore patient recruitment is to low
Sponsor: University Hospital Muenster (Other)
Collaborators: International Anesthesia Research Society (IARS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-AnIt-06
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Elective Surgical Procedure; Colorectal Surgery
Keywords: Systemic lidocaine; peridural lidocaine; perioperative analgesia; inflammation; Anesthesia
MeSH Terms: conditions — Inflammation | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Lidocaine i.v
  Interventions: Drug: lidocaine
- 2 (Active Comparator): intraoperatively lidocaine epidural postoperatively lidocaine i.v.
  Interventions: Drug: lidocaine
- 3 (Active Comparator): intraoperatively lidocaine i.v. postoperatively lidocaine epidural
  Interventions: Drug: lidocaine
- 4 (Active Comparator): lidocaine epidural
  Interventions: Drug: lidocaine
- 5 (Placebo Comparator): placebo i.v.
  Interventions: Drug: NaCl 0,9%

INTERVENTIONS:
Drug: lidocaine — administration of lidocaine intravenously or epidural or administration of placebo
  Arms: 1; 2; 3; 4
Drug: NaCl 0,9% — Administration of placebo i.v.
  Arms: 5

SUMMARY:
The purpose of this study is to comparing effects of intravenously (IV) administered lidocaine to effects of epidurally (ED) administered lidocaine in patients undergoing elective colorectal surgery

ELIGIBILITY:
Inclusion Criteria:

* elective colorectal surgery

Exclusion Criteria:

* ASA > 3
* history of anti-inflammatory therapy
* history of inflammatory bowl diseases
* history of chronic pain treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-09; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
length of postoperative hospital stay | end of hospital stay

SECONDARY OUTCOMES:
Hyperalgesia perioperative | postoperative day 2, 4, 8, end of hospital stay and follow-up
Cytokine levels perioperative | before surgery and 4 hours, 2 and 4 days after surgery
Bowel motility perioperative | days after surgery
Length of PACU stay | end of PACU stay
Cognitive function perioperatively | before surgery, one and four days after surgery, at end of hospital stay and follow-up
Incidence of wound healing disturbances | within 4 weeks after surgery
Postoperative Analgesia | until end of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: K Hahnenkamp, MD, Study Chair — Department of Anesthesiology and Intensive Care, University Hospital Muenster
Locations (3):
- Germany (3):
  - University Hospital Muenster, Münster
  - St. Franziskushospital Muenster, Münster
  - St. Marienhospital, Vechta

REFERENCES:
- [Background] Kuo CP, Jao SW, Chen KM, Wong CS, Yeh CC, Sheen MJ, Wu CT. Comparison of the effects of thoracic epidural analgesia and i.v. infusion with lidocaine on cytokine response, postoperative pain and bowel function in patients undergoing colonic surgery. Br J Anaesth. 2006 Nov;97(5):640-6. doi: 10.1093/bja/ael217. Epub 2006 Sep 4. PMID 16952918
- [Background] Cooke ED, Bowcock SA, Lloyd MJ, Pilcher MF. Intravenous lignocaine in prevention of deep venous thrombosis after elective hip surgery. Lancet. 1977 Oct 15;2(8042):797-9. doi: 10.1016/s0140-6736(77)90727-9. PMID 71604